CLINICAL TRIAL: NCT06596889
Title: The Effect of Assistive Airway Equipment on Intubation-Related Events in the Perioperative Period
Brief Title: The Effect of Assistive Airway Equipment on Intubation
Status: Active, not recruiting | Type: Observational
Sponsor: Kocaeli City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024-87
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Airway Management; Airway Complication of Anaesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Not any equipment: Control group
  Interventions: Procedure: Successful airway management
- Other types of equipment: Brand new oral airways
  Interventions: Procedure: Successful airway management

INTERVENTIONS:
Procedure: Successful airway management — * Types of equipment: Traditional oral airways, new airways, etc.
  * Professional experience of the airway management practitioner (in years).
  * If advanced, type of airway complication (bleeding, dental damage, mucosal damage, etc.), number of attempts
  will be recorded separately for each patient.

SUMMARY:
In this study, investigators will research the types and incidence rates of airway complications seen in the perioperative period during airway management. In addition, unlike the literature, the relationship between the airway equipment used and perioperative airway complications will be investigated.

DETAILED DESCRIPTION:
Complications related to airway management rarely occur in the operating room; however, these complications can lead to life-threatening situations. There are many studies on the types and incidence rates of airway management complications in the perioperative period. However, although the types and incidence rates of airway complications have been investigated in these studies, the effect of airway equipment used in airway management on complications has not been investigated. There are many equipment used in airway management. Laryngoscopes, face masks, oral airway devices and many assistant airway management devices are used as basic equipment. Different airway equipment may be used in each center in each case. There is no standard between centers in this regard.

In this study, investigators will primarily research the types and incidence rates of airway complications seen in the perioperative period during airway management similar to the existing literature. In addition, unlike the literature, the relationship between the airway equipment used and perioperative airway complications will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 18 and 75.
2. Patients who will undergo elective surgery.
3. Patients to be operated under general anesthesia.
4. Patients without difficult airway markers

Exclusion Criteria:

1. Patients to be operated with emergency surgical indication.
2. Patients to be operated with regional anesthesia.
3. Patients with expected difficult airway markers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study was prospective and observational. There is no grouping. Oral and written informed consent will be obtained from the patients in the preoperative ward or in the preoperative preparation room of the operating room.
  Patients scheduled for elective operation under general anesthesia whose consents were obtained will be included in the study. Airway management techniques and equipment used will not be interfered with.
  After the patient's airway management is completed: the following data will be recorded.
  * Types of equipment: laryngoscopes, face masks, oral airways, styli, plugs, etc.
  * Professional experience of the airway management practitioner (in years).
  * If advanced, type of airway complication (bleeding, dental damage, mucosal damage, etc.), number of attempts.
Sampling Method: Non-Probability Sample
Enrollment: 870 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
The incidence of airway complications seen in the induction of anesthesia. | The first 15 minutes during induction of anesthesia
  The incidence of complications (mucosal bleeding, tooth damage, etc.) that may occur during induction of anesthesia with different airway devices will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Yılmaz, Principal Investigator — Kocaeli City Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Kocaeli City Hospital, Kocaeli
  - University of Health Sciences Sanliurfa Mehmet Akif Inan Training and Research Hospital, Sanliurfa

IPD SHARING:
Plan to Share IPD: No